CLINICAL TRIAL: NCT03884634
Title: Efficacy of the Dabir Surfaces Micropressure Overlay for Decubitus Ulcer Prevention During Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Eric Roselli, M. D., Principal Investigator, The Cleveland Clinic
Other Study IDs: 18-928
Record Dates: First submitted 2019-02-20; First posted 2019-03-21 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Pressure Ulcer; Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dabir Microsurface Overlay Group: Patients undergoing cardiac surgery with the Dabir Micropressure Overlay in place and turned ON (in addition to standard operating room table mattress and heating/cooling gel pad).
  Interventions: Device: Dabir Micropressure Overlay
- Control Group: Patients undergoing cardiac surgery with the Dabir Micropressure Overlay in place and turned OFF (in addition to standard operating room table mattress and heating/cooling gel pad).

INTERVENTIONS:
Device: Dabir Micropressure Overlay — The study intervention is the use of the Dabir micropressure overlay on the operating room table during surgical operations. The device is positioned on top of a standard foam pad and gel heat exchanger. The overlay is already in use in some (but not all) adult cardiac operating rooms.
  The overlay will be present on the operating room table for all adult cardiac operations. On odd calendar dates the device will be powered on, and on even calendar dates the device will be powered off.
  Groups: Dabir Microsurface Overlay Group

SUMMARY:
This is a systematic random sampling study of the effects of the Dabir Micropressure Overlay on perioperative pressure injuries during cardiac surgery.

DETAILED DESCRIPTION:
This is a simple pragmatic systematic quality improvement study aimed at real-world evaluation of a device claimed to reduce pressure ulcers in patients undergoing cardiac surgery.

Data acquisition will be based on systematic sampling of cardiac surgery operations based on odd and even calendar dates. On odd dates the Dabir micropressure overlay will be functional on the operating room tables. On even dates the Dabir micropressure overlay will not be functional on the operating room tables. Data on baseline characteristics, operative parameters, and primary and secondary endpoints will be gathered from STS and wound care sources, which are routinely collected for all patients. There will be no additional patient information and data collected specifically for this study.

ELIGIBILITY:
Inclusion Criteria:

* All cases scheduled in the cardiac surgery OR suites at the CCF main campus.

Exclusion Criteria:

* Patients who have had previous surgery within 5 days of enrollment in the study will excluded from analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be all adult patients undergoing cardiac surgery at Cleveland Clinic main campus during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 6627 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Number of patient developing new perioperative pressure ulcers | 5 days from operation
  New pressure ulcers, any stage

SECONDARY OUTCOMES:
Pressure ulcer stage | 5 day from operation
  Pressure ulcer stage, according to NPUAP staging system
Number of wound care consultations | From date of surgery until 30 days or the date of hospital discharge or the date of death from any cause, whichever came first, assessed up to 3 months
  How often patients require consultation by the specialized wound care team for assessment and treatment of skin issues

CONTACTS AND LOCATIONS:
Overall Officials: Eric Roselli, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No